CLINICAL TRIAL: NCT00583076
Title: A Pilot Study of the Safety and Efficacy of AST-120 in the Treatment of Active Pouchitis
Brief Title: Safety and Efficacy of AST-120 in the Treatment of Pouchitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-908
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Pouchitis
Keywords: Pouchitis; Active Pouchitis; Safety and Efficacy of AST120
MeSH Terms: conditions — Pouchitis | interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AST-120, 2grams, three times daily
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — AST-120, 2grams,three times daily for 4 weeks. Responders in the second cohort of patients are eligible to receive AST-120 for up to 52 weeks.

SUMMARY:
The aim of the study is to assess the safety and efficacy of an investigational agent, AST-120, in treating patients with active pouchitis. This is an open-label trial which means that all patients will receive AST-120 in 2g sachets (packets)three times a day for 4 weeks. All antibiotics, probiotics and nutritional agents must have been discontinued for at least 2 weeks prior to study entry. An initial group of 10 patients will be enrolled. If there are no serious adverse events associated with the study drug and at least 3 of the 10 patients respond, a second group of 10 patients will be enrolled. In the second group of patients, those patients who are considered responders or who are in remission are eligible to receive open-label AST-120 for as long as response is maintained up to a maximum of 52 weeks. Patients will have clinic visits at the start of the study and at week 4. If continuing on open label AST-120 after week 4, patients will have clinic visits every 12 weeks to assess the continuing safety and efficacy of AST-120. Endoscopies will be performed at the start of the study, week 4, week 28, week 52 or early termination.

DETAILED DESCRIPTION:
The management and prognosis vary in different types of pouchitis. For antibiotic-responsive pouchitis, the first-line therapy includes a 2-week course of metronidazole or ciprofloxacin. A relapsing course of pouchitis is common. Of the patients with acute pouchitis, 61% would develop at least one recurrence. Typically, patient's symptoms and endoscopic and histologic inflammation respond favorably to antibiotic therapy, but symptoms quickly recur when antibiotics are discontinued. This group of patients is classified as having antibiotic-dependent pouchitis and often requires long-term antibiotic or probiotic therapy to keep the disease in remission.

Although the majority of patients with active pouchitis respond favorably to antibiotic therapy, relapse is common, which often requires frequent antibiotic therapy. The concerns about frequent use of antibiotic agents are: 1)antibiotics such as metronidazole often cause adverse effects; 2)long-term or frequent use of antibiotics, including ciprofloxacin, metronidazole, and rifaximin, often leads to bacterial resistance. In clinical practice, we have encountered more and more patients with antibiotic-refractory pouchitis, which could largely be due to overuse of antibiotic agents; 3)UC patients with IPAA have an increased risk for the development of intra-abdominal infections, such as pouch leaks, abscess, and cholangitis from primary sclerosing cholangitis, which require antibiotic therapy with agents similar to the agents used in pouchitis. Bacterial resistance developed from the overuse of antibiotics for pouchitis might jeopardize the treatment of other intra-abdominal infections; 4) overuse of antibiotics can lead to overload of certain commensal bacteria or pathogenic bacteria, leading to pouch inflammation. Therefore, safe and effective agents are needed to treat active pouchitis, particularly on a long-term basis.

AST-120 is manufactured by Kureha Corporation, Japan. The agent was approved in Japan in 1992 for the treatment of patients with chronic kidney disease (CKD). It is comprised of highly adsorptive, porous, spherical carbon particles and is packaged in 2 g sachets for oral administration designed for the treatment of gastrointestinal diseases. AST-120 consists of black microspheres approximately 0.2-0.4 mm in diameter with high adsorption ability and large surface area. Composed mainly of carbon (approximately 96%), the clinical utility of AST-120 is thought to reside in its ability to adsorb low molecular weight toxins, inflammatory mediators, and harmful bile acid products from the gastrointestinal tract, preventing local toxicity and their systemic absorption. AST-120 has a selective adsorption profile for certain acidic and basic organic compounds, and has a significantly lower adsorptive capacity than activated charcoal for digestive enzymes.

This study is an open-label pilot trial in which all patients will receive AST-120 in 2 g sachets three times a day (to be taken between meals at 10:00 am, 3:00 pm, and immediately before going to bed) for 4 complete weeks. AST-120 is a tasteless, odorless, oral preparation. To take the product, patients will tear open the sachets, drop the contents directly on their tongue and wash it down with 8 ounces of water. All antibiotics, probiotics and nutritional agents must have been discontinued for at least 2 weeks prior to study entry. For purposes of this trial response is defined as a > or = 3 point reduction in the 18-point PDAI scoring system. Remission is defined as a PDAI score < 7.

The study population will consist of patients with active pouchitis after ileal pouch-anal anastomosis for Ulcerative Colitis (UC) present with primary symptoms such as increased stool frequency and abdominal pain. The diagnosis of active pouchitis will be defined by a PDAI score > 7 points, with a combined assessment of symptoms, endoscopy, and histology.

An initial cohort of 10 patients will be enrolled. Based on the efficacy outcome (at least 3 out of 10 patients responding) and safety outcome (no significant adverse event associated with study drug) a second cohort of 10 patients will be treated. Patients in the second cohort who are considered responders (i.e., have had at least a 3 point reduction in the 18 point PDAI scoring system) or who are in remission (PDAI<7) are eligible to receive open-label AST-120 for as long as response is maintained up to a maximum of 52 weeks. If, at any time, the patient relapses (PDAI>7 for patients who were in remission, or an increase in PDAI such that at least a 3 point reduction is not maintained for responders), open-label treatment will be discontinued and the patient will be removed from the study. Patients will also discontinue open-label treatment and be removed from the study if warranted by treatment-emergent safety concerns or if, in the opinion of the investigator, it is in the patient's best interest to discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a current episode of active pouchitis (defined as having a PDAI score > 7) after IPAA for UC confirmed by endoscopy and histology
* Patients with active pouchitis who have never been treated with antibiotics (antibiotic-naive) or who have been previously treated with antibiotics and responded. Antibiotic-dependent patients may be enrolled as long as antibiotic use is discontinued for at least two weeks prior to study entry. Antibiotic-dependent pouchitis is defined as a condition in which a patient with frequent episodes (> or = 4 episodes per year) of pouchitis or persistent symptoms requires long-term, continuous antibiotic or probiotic therapy to keep the disease in remission.
* Able to give informed consent
* Able and willing to comply with all study procedures
* Females must be post-menopausal, surgically incapable of bearing children, or practicing a reliable single barrier method of birth control (condom, intrauterine devices, spermicide and barrier, Depot). Partner/spouse sterility may also qualify at the investigator's discretion. Females of child-bearing potential must have a negative urine pregnancy test at baseline. Oral contraceptives are not acceptable as there is a potential interaction with AST-120.

Exclusion Criteria:

* Patients previously treated with infliximab or any investigational immunosuppressant/immunomodulator
* Patients whose condition is severe enough that, in the investigator's opinion, withholding antibiotics for 4 weeks during the AST-120 trial is not feasible
* Patients undergoing chemotherapy for the treatment of cancer
* Antibiotic use within 2 weeks prior to the entry of the study
* Crohn's disease of the pouch, including inflammatory, fibrostenotic, or fistulizing phenotypes, based on the previously established diagnostic criteria (Shen B, et al. Am J Gastroenterol 2006 in press)
* Active specific infection of the pouch: cytomegalovirus infection and C. difficile infection
* Patients with chronic antibiotic-refractory pouchitis. Antibiotic- refractory pouchitis is defined as a condition where a patient fails to respond to a 4 week course of a single antibiotic (metronidazole or ciprofloxacin), requiring prolonged therapy of > or = 4 weeks consisting of 2 antibiotics, oral or topical 5-aminosalicylate, corticosteroid therapy, or oral immunomodulator therapy.
* History of non-inflammatory disease of the pouch: decreased pouch compliance, irritable pouch syndrome, afferent or efferent limb obstruction
* Isolated cuffitis. Patients who have active pouchitis as the predominant condition, but also have cuffitis may be enrolled.
* Strictures of the pouch inlet or outlet
* Ileal pouch patients with familial adenomatous polyposis
* History of lactose intolerance
* Known celiac disease
* Primary sclerosing cholangitis (PSC) with or without liver transplant; PSC with or without Actigall or Urso therapy
* Uncontrolled systemic diseases
* Needing oral or topical steroid treatment or 5-ASA agents
* Other major physical or major psychiatric illness within the last 6 months that in the opinion of the investigator would affect the patient's ability to complete the trial
* Active use of cholestyramine
* Active use of NSAIDs or aspirin
* Women who are pregnant, breast feeding, or planning to become pregnant during the study
* Patients who are on therapy of 5-ASA at the entry of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Remission induction as defined by a Pouchitis Disease Activity Index (PDAI) score < 7 (Sandborn et al, Mayo Clin Proc 1994), as well as maintenance of remission over 12 months | 4 weeks induction, 12 months maintenance of remission
Safety: Any adverse events (AEs) deemed possibly, probably, or definitely related to treatment with investigational product | 4 weeks induction, 12 months maintenance of remission

SECONDARY OUTCOMES:
Response defined as a > or = 3 point reduction in the 18-point PDAI scoring system | 4 weeks, weeks 28 and 52
Reduction of PDAI clinical symptom score, range from 0 to 6 (e.g., stoll frequency returns to the normal baseline) | 4 weeks, weeks 28 and 52
Reduction of PDAI endoscopic score, range from 0 to 6 | 4 weeks, weeks 28 and 52
Reduction of PDAI histology score, range from 0 to 6 | 4 weeks, weeks 28 and 52
Need for rescue medication or increased quantity of antidiarrheal medication used during the trial | 4 weeks, weeks 28 and 52
Quality of Life (Cleveland Global Quality of Life [CGQL] and Short Inflammatory Bowel Disease Questionnaire [SIBDQ] | 4 weeks, through 52 weeks
Clinical laboratory tests including liver transaminases and alkaline phosphatase | 4 weeks, through 52 weeks
Worsening GI symptoms (diarrhea, abdominal pain, urgency or bleeding) or new GI and ex-intestinal systemic symptoms (such as headache, nausea, vomiting, and constipation) | 4 weeks, through 52 weeks
Physical examination, vital signs (blood pressure, heart rate, respiration rate and temperature) | 4 weeks, through 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bo Shen, MD, Principal Investigator — Clevland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Loftus EV Jr, Silverstein MD, Sandborn WJ, Tremaine WJ, Harmsen WS, Zinsmeister AR. Ulcerative colitis in Olmsted County, Minnesota, 1940-1993: incidence, prevalence, and survival. Gut. 2000 Mar;46(3):336-43. doi: 10.1136/gut.46.3.336. PMID 10673294
- [Background] Dhillon S; Loftus EV; Tremaine WJ; Jewell DA; Harmsen WS; Zinsmeister AR; Melton LJ; Pemberton H; Wolff BG; Dozois EJ; Cima RR; Larson DW; Sandborn WJ. The natural history of surgery for ulcerative colitis in a population based cohort from Olmsted County, Minnesota. Am J Gastroenterol 2005;100:A819
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Penna C, Dozois R, Tremaine W, Sandborn W, LaRusso N, Schleck C, Ilstrup D. Pouchitis after ileal pouch-anal anastomosis for ulcerative colitis occurs with increased frequency in patients with associated primary sclerosing cholangitis. Gut. 1996 Feb;38(2):234-9. doi: 10.1136/gut.38.2.234. PMID 8801203
- [Background] Fazio VW, Ziv Y, Church JM, Oakley JR, Lavery IC, Milsom JW, Schroeder TK. Ileal pouch-anal anastomoses complications and function in 1005 patients. Ann Surg. 1995 Aug;222(2):120-7. doi: 10.1097/00000658-199508000-00003. PMID 7639579
- [Background] Penna C, Tiret E, Kartheuser A, Hannoun L, Nordlinger B, Parc R. Function of ileal J pouch-anal anastomosis in patients with familial adenomatous polyposis. Br J Surg. 1993 Jun;80(6):765-7. doi: 10.1002/bjs.1800800638. PMID 8392425
- [Background] Tjandra JJ, Fazio VW, Church JM, Oakley JR, Milsom JW, Lavery IC. Similar functional results after restorative proctocolectomy in patients with familial adenomatous polyposis and mucosal ulcerative colitis. Am J Surg. 1993 Mar;165(3):322-5. doi: 10.1016/s0002-9610(05)80834-7. PMID 8383471
- [Background] Carter MJ, Di Giovine FS, Cox A, Goodfellow P, Jones S, Shorthouse AJ, Duff GW, Lobo AJ. The interleukin 1 receptor antagonist gene allele 2 as a predictor of pouchitis following colectomy and IPAA in ulcerative colitis. Gastroenterology. 2001 Oct;121(4):805-11. doi: 10.1053/gast.2001.28017. PMID 11606494
- [Background] Brett PM, Yasuda N, Yiannakou JY, Herbst F, Ellis HJ, Vaughan R, Nicholls RJ, Ciclitira PJ. Genetic and immunological markers in pouchitis. Eur J Gastroenterol Hepatol. 1996 Oct;8(10):951-5. doi: 10.1097/00042737-199610000-00003. PMID 8930557
- [Background] Meier CB, Hegazi RA, Aisenberg J, Legnani PE, Nilubol N, Cobrin GM, Duerr RH, Gorfine SR, Bauer JJ, Sachar DB, Plevy SE. Innate immune receptor genetic polymorphisms in pouchitis: is CARD15 a susceptibility factor? Inflamm Bowel Dis. 2005 Nov;11(11):965-71. doi: 10.1097/01.mib.0000186407.25694.cf. PMID 16239841
- [Background] Sandborn WJ. Pouchitis following ileal pouch-anal anastomosis: definition, pathogenesis, and treatment. Gastroenterology. 1994 Dec;107(6):1856-60. doi: 10.1016/0016-5085(94)90832-x. No abstract available. PMID 7958702
- [Background] Duffy M, O'Mahony L, Coffey JC, Collins JK, Shanahan F, Redmond HP, Kirwan WO. Sulfate-reducing bacteria colonize pouches formed for ulcerative colitis but not for familial adenomatous polyposis. Dis Colon Rectum. 2002 Mar;45(3):384-8. doi: 10.1007/s10350-004-6187-z. PMID 12068199
- [Background] Nasmyth DG, Godwin PG, Dixon MF, Williams NS, Johnston D. Ileal ecology after pouch-anal anastomosis or ileostomy. A study of mucosal morphology, fecal bacteriology, fecal volatile fatty acids, and their interrelationship. Gastroenterology. 1989 Mar;96(3):817-24. PMID 2914643
- [Background] Gosselink MP, Schouten WR, van Lieshout LM, Hop WC, Laman JD, Ruseler-van Embden JG. Eradication of pathogenic bacteria and restoration of normal pouch flora: comparison of metronidazole and ciprofloxacin in the treatment of pouchitis. Dis Colon Rectum. 2004 Sep;47(9):1519-25. doi: 10.1007/s10350-004-0623-y. Epub 2004 Jul 8. PMID 15486751
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Brzezinski A, Bevins CL, Bambrick ML, Seidner DL, Fazio VW. A randomized clinical trial of ciprofloxacin and metronidazole to treat acute pouchitis. Inflamm Bowel Dis. 2001 Nov;7(4):301-5. doi: 10.1097/00054725-200111000-00004. PMID 11720319
- [Background] Shen B, Fazio VW, Remzi FH, Bennett AE, Lopez R, Brzezinski A, Oikonomou I, Sherman KK, Lashner BA. Combined ciprofloxacin and tinidazole therapy in the treatment of chronic refractory pouchitis. Dis Colon Rectum. 2007 Apr;50(4):498-508. doi: 10.1007/s10350-006-0828-3. PMID 17279300
- [Background] Ohge H, Furne JK, Springfield J, Rothenberger DA, Madoff RD, Levitt MD. Association between fecal hydrogen sulfide production and pouchitis. Dis Colon Rectum. 2005 Mar;48(3):469-75. doi: 10.1007/s10350-004-0820-8. PMID 15747080
- [Background] Smith FM, Coffey JC, Kell MR, O'Sullivan M, Redmond HP, Kirwan WO. A characterization of anaerobic colonization and associated mucosal adaptations in the undiseased ileal pouch. Colorectal Dis. 2005 Nov;7(6):563-70. doi: 10.1111/j.1463-1318.2005.00833.x. PMID 16232236
- [Background] Kmiot WA, Youngs D, Tudor R, Thompson H, Keighley MR. Mucosal morphology, cell proliferation and faecal bacteriology in acute pouchitis. Br J Surg. 1993 Nov;80(11):1445-9. doi: 10.1002/bjs.1800801132. PMID 8252361
- [Background] Gionchetti P, Rizzello F, Venturi A, Ugolini F, Rossi M, Brigidi P, Johansson R, Ferrieri A, Poggioli G, Campieri M. Antibiotic combination therapy in patients with chronic, treatment-resistant pouchitis. Aliment Pharmacol Ther. 1999 Jun;13(6):713-8. doi: 10.1046/j.1365-2036.1999.00553.x. PMID 10383499
- [Background] Shen B, Goldblum JR, Hull TL, Remzi FH, Bennett AE, Fazio VW. Clostridium difficile-associated pouchitis. Dig Dis Sci. 2006 Dec;51(12):2361-4. doi: 10.1007/s10620-006-9172-7. Epub 2006 Nov 11. PMID 17103037
- [Background] Shen BO, Jiang ZD, Fazio VW, Remzi FH, Rodriguez L, Bennett AE, Lopez R, Queener E, Dupont HL. Clostridium difficile infection in patients with ileal pouch-anal anastomosis. Clin Gastroenterol Hepatol. 2008 Jul;6(7):782-8. doi: 10.1016/j.cgh.2008.02.021. Epub 2008 May 7. PMID 18467184
- [Background] Natori H, Utsunomiya J, Yamamura T, Benno Y, Uchida K. Fecal and stomal bile acid composition after ileostomy or ileoanal anastomosis in patients with chronic ulcerative colitis and adenomatosis coli. Gastroenterology. 1992 Apr;102(4 Pt 1):1278-88. PMID 1312975
- [Background] Salemans JM, Nagengast FM. Clinical and physiological aspects of ileal pouch-anal anastomosis. Scand J Gastroenterol Suppl. 1995;212:3-12. doi: 10.3109/00365529509090295. PMID 8578229
- [Background] Nasmyth DG, Johnston D, Williams NS, King RF, Burkinshaw L, Brooks K. Changes in the absorption of bile acids after total colectomy in patients with an ileostomy or pouch-anal anastomosis. Dis Colon Rectum. 1989 Mar;32(3):230-4. doi: 10.1007/BF02554535. PMID 2493363
- [Background] Lerch MM, Braun J, Harder M, Hofstadter F, Schumpelick V, Matern S. Postoperative adaptation of the small intestine after total colectomy and J-pouch-anal anastomosis. Dis Colon Rectum. 1989 Jul;32(7):600-8. doi: 10.1007/BF02554181. PMID 2737061
- [Background] de Silva HJ, Millard PR, Kettlewell M, Mortensen NJ, Prince C, Jewell DP. Mucosal characteristics of pelvic ileal pouches. Gut. 1991 Jan;32(1):61-5. doi: 10.1136/gut.32.1.61. PMID 1846839
- [Background] Sauser P; Fitsher A; Riedel HD; Kleiner H; Kramer W; Stengelin S; Stremmel W; Stiehl A. Reduced transcription of ileal bile acid transporters during chronic ileal inflammation in man. Gastroenterol 2000;118:A4296
- [Background] Levitt MD, Kuan M. The physiology of ileo-anal pouch function. Am J Surg. 1998 Oct;176(4):384-9. doi: 10.1016/s0002-9610(98)00194-9. PMID 9817261
- [Background] Breuer NF, Rampton DS, Tammar A, Murphy GM, Dowling RH. Effect of colonic perfusion with sulfated and nonsulfated bile acids on mucosal structure and function in the rat. Gastroenterology. 1983 May;84(5 Pt 1):969-77. PMID 6299874
- [Background] Merrett MN; Crotty BJ; Mortensen N; Jewell DP. Ileal pouch dialysate is cytotoxic to I-407 and HT-29 cells: Bile may be the active factor. Gut 1991;32:A1205
- [Background] Shen B, Fazio VW, Remzi FH, Delaney CP, Bennett AE, Achkar JP, Brzezinski A, Khandwala F, Liu W, Bambrick ML, Bast J, Lashner B. Comprehensive evaluation of inflammatory and noninflammatory sequelae of ileal pouch-anal anastomoses. Am J Gastroenterol. 2005 Jan;100(1):93-101. doi: 10.1111/j.1572-0241.2005.40778.x. PMID 15654787
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Bevins CL, Brzezinski A, Petras RE, Fazio VW. Endoscopic and histologic evaluation together with symptom assessment are required to diagnose pouchitis. Gastroenterology. 2001 Aug;121(2):261-7. doi: 10.1053/gast.2001.26290. PMID 11487535
- [Background] Moskowitz RL, Shepherd NA, Nicholls RJ. An assessment of inflammation in the reservoir after restorative proctocolectomy with ileoanal ileal reservoir. Int J Colorectal Dis. 1986 Jul;1(3):167-74. doi: 10.1007/BF01648445. PMID 3039030
- [Background] Sandborn WJ, Tremaine WJ, Batts KP, Pemberton JH, Phillips SF. Pouchitis after ileal pouch-anal anastomosis: a Pouchitis Disease Activity Index. Mayo Clin Proc. 1994 May;69(5):409-15. doi: 10.1016/s0025-6196(12)61634-6. PMID 8170189
- [Background] Sandborn WJ. Pouchitis: Risk factors, frequency, natural history, classification and public health prospective. In: McLead R; Martin F; Sutherland L; Wallace J; Williams C, eds. Trends in Inflammatory Bowel Disease 1996. Lancaster UK: Kluwer Academic Publishers, 1997:51-63
- [Background] Shen B. Diagnosis and treatment of patients with pouchitis. Drugs. 2003;63(5):453-61. doi: 10.2165/00003495-200363050-00002. PMID 12600225
- [Background] Zuccaro G Jr, Fazio VW, Church JM, Lavery IC, Ruderman WB, Farmer RG. Pouch ileitis. Dig Dis Sci. 1989 Oct;34(10):1505-10. doi: 10.1007/BF01537101. PMID 2791801
- [Background] Lohmuller JL, Pemberton JH, Dozois RR, Ilstrup D, van Heerden J. Pouchitis and extraintestinal manifestations of inflammatory bowel disease after ileal pouch-anal anastomosis. Ann Surg. 1990 May;211(5):622-7; discussion 627-9. PMID 2339922
- [Background] Shen B, Fazio VW, Remzi FH, Brzezinski A, Bennett AE, Lopez R, Hammel JP, Achkar JP, Bevins CL, Lavery IC, Strong SA, Delaney CP, Liu W, Bambrick ML, Sherman KK, Lashner BA. Risk factors for diseases of ileal pouch-anal anastomosis after restorative proctocolectomy for ulcerative colitis. Clin Gastroenterol Hepatol. 2006 Jan;4(1):81-9; quiz 2-3. doi: 10.1016/j.cgh.2005.10.004. PMID 16431309